CLINICAL TRIAL: NCT02727140
Title: Yoga as a Supportive Therapy for Patients With Hypertension: A Randomized Controlled Trial
Brief Title: Yoga as a Supportive Therapy for Patients With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Holger Cramer, Research director, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15-6726-BO
Record Dates: First submitted 2016-03-23; First posted 2016-04-04 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Yoga

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Yoga with Asana (yoga postures) (Experimental)
  Interventions: Behavioral: Yoga with Asana (yoga postures)
- Yoga without Asana (yoga postures) (Experimental)
  Interventions: Behavioral: Yoga without Asana (yoga postures)
- Wait-list control group (No Intervention)

INTERVENTIONS:
Behavioral: Yoga with Asana (yoga postures) — Yoga intervention consisting of asana, breathing and relaxation, meditation
  Arms: Yoga with Asana (yoga postures)
Behavioral: Yoga without Asana (yoga postures) — Yoga intervention without asanas, consisting only of breathing, relaxation and meditation
  Arms: Yoga without Asana (yoga postures)

SUMMARY:
The proposed study aims to investigate the feasibility, effectiveness, and perceived benefit of a supportive hatha yoga intervention for patients with hypertension using antihypertensive drugs. Patients will be randomized into 3 groups comparing hatha yoga with yoga postures, breathing and relaxation techniques to a hatha yoga intervention without yoga postures (only breathing and relaxation techniques) as well as to a wait list control group.

ELIGIBILITY:
Inclusion Criteria:

* essential Hypertension
* stable antihypertensive medication during the next 6 months

Exclusion Criteria:

* pregnancy or breast feeding
* simultaneous participation in further clinical intervention trials
* regular yoga practice in the past 12 months
* serious mental illness (severe depression, severe addiction, psychosis)
* manifest coronary heart disease that has been treated in the past 3 months or myocardial infarction, embolism of pulmonary arteries or stroke in the past 3 months
* heart failure ≥ state 1 New York Heart Association (NYHA)
* peripheral arterial occlusive disease ≥ state 1
* renal insufficiency > state 2, glomerular filtration rate < 60 ml/min/1,73m² according to he National Kidney Foundation (NKF)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
24 h mean value of systolic and diastolic blood pressure | 12 weeks

SECONDARY OUTCOMES:
24 h mean value of systolic and diastolic blood pressure | 28 weeks
Health-related Quality of Life | 12 weeks
  Short Form 36 Health Survey Questionnaire (SF-36)
Health-related Quality of Life | 28 weeks
  Short Form 36 Health Survey Questionnaire (SF-36)
Emotional Distress | 12 weeks
  Hospital Anxiety and Depression Scale (HADS)
Emotional Distress | 28 weeks
  Hospital Anxiety and Depression Scale (HADS)
Subjective Stress | 12 weeks
  Cohen Perceived Stress Scale (CPSS)
Subjective Stress | 28 weeks
  Cohen Perceived Stress Scale (CPSS)
Nutrition habits | 12 weeks
  Five a Day Food Frequency Questionnaire
Nutrition habits | 28 weeks
  Five a Day Food Frequency Questionnaire
Physical activity | 12 weeks
  Baecke Physical Activity Questionnaire
Physical activity | 28 weeks
  Baecke Physical Activity Questionnaire
Adverse Events | 12 weeks
Adverse Events | 28 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal and Integrative Medicine, Kliniken Essen-Mitte, Essen, Germany

IPD SHARING:
Plan to Share IPD: No